CLINICAL TRIAL: NCT07162831
Title: Metacognitive Intervention in Children and Adolescents With ADHD - MiA Study
Acronym: MiA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BASEC2025-01189
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: ADHD
Keywords: Metacognition; ADHD; Cognitive training; Children; Adolescents; Cognitive development
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): Training with Mio-Training for 5 weeks, three times per week.
  Interventions: Behavioral: Mio-Training
- Control group (No Intervention): Waiting control group. Participants may use the Mio-Training after completion of the last follow-up assessment.

INTERVENTIONS:
Behavioral: Mio-Training — The Mio-Training aims to increase metacognitive knowledge, teaches mnemonic skills, trains the working memory capacity and coordinative skills to strenghten cognitive development in children and adolescents with ADHD.
  Arms: Training group

SUMMARY:
The aim of the MiA-Study is to address the current lack of effective treatment options to reduce cognitive and physical long-term problems in children and adolescents with Attention Deficit Hyperactivity Disorder (ADHD). Through the use of the Mio-Training, cognitive development will be strengthened and metacognitive thinking and awareness will increase.

The MiA-Study is conducted additionally to the Mio-study to evaluate the effectiveness of the Mio-Training specifically within the ADHD population.

The Mio-Training for children and adolescence with ADHD includes a combination of cognitive and coordinative training tasks and prospective as well as retrospective metacognitive questions. In a randomized controlled trial, the Mio-Training will be analysed for its efficacy on metacognitive thinking and executive functions. In particular, the investigators are interested in factors that affect the efficacy of the training program such as compliance, age, sex or the severity of the ADHD. This study will give insight into the role of metacognition in cognitive performance and will foster the development of children and adolescents with ADHD in the long-term.

DETAILED DESCRIPTION:
In the MiA-Study, the investigators investigate a newly developed Training program at the interface between neuropsychology and sports science - the Mio-Training - for its efficacy. The aim of the Mio-Training is to strengthen the cognitive development of children and adolescents with ADHD in the long-term. The Mio-Training contains a combination of cognitive and coordinative training tasks and metacognitive questions to promote knowledge and awareness of one's own thinking. In order to counteract the shortage of skilled workers and the increasing specialization of individual specialist areas, solutions are needed that can be implemented without a lot of staff. From today's perspective, there are hardly any trainings for children and adolescents that show long-term effects on cognitive development and can also be transferred to non-trained tasks in school and everyday life.

The investigators are testing the effectiveness of the Mio-Training in a randomized clinical trial (RCT) and expect a strengthening of metacognition and core cognitive functions (i.e. executive functions). The MiA-Study will provide information about the role of metacognition in cognitive performance and, ideally, provide evidence for a novel, interdisciplinary rehabilitation strategy for children and adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (see Informed Consent Form) of participants and / or one parent / legal guardian
* Age 8-16 years
* A diagnosis of ADHD (mild, moderate or severe)
* Intelligence >85 (WISC-V short form)
* German or french speaking
* Willingness to perform the assessments without the medication (the study visits will take place without ADHD medication)

Exclusion Criteria:

* Any other instable neurological condition (e.g. epilepsy) that significantly impairs development
* A severe psychiatric disease (e.g., eating disorder) or severe learning disability that significantly impairs development
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Junior Metacognitive Awareness Inventory (Jr.MAI) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up
  Total score of the Junior Metacognitive Awareness Inventory over the three timepoints (baseline, immediate followup & 3-months follow-up). Raw values ranging 18-90. Higher scores mean better outcome.

SECONDARY OUTCOMES:
Wechsler Intelligence Scale For Children: 5th Ed (WISC-V) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Indices ranging from 0 to 155. Higher scores mean better outcome.
Color-Word Interference Test (Delis-Kaplan Executive Function System; D-KEFS) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Scaled Scores ranging from 1 to 19. Higher scores mean better outcome.
Tower of Hanoi (D-KEFS) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Scaled Scores ranging from 1 to 19. Higher scores mean better outcome.
Verbal learning and memory test (VLMT) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.
Pattern learning (Memory and Learning Test; Basic-MLT) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.
Test Battery for Attention Assessment (TAP) | At baseline; immediately (up to 1 week) after the training or waiting period.
  T-scores ranging from 20 to 80 (M = 50, SD = 10). Higher scores mean better outcome.
German Motor Performance Test (DMT) | At baseline; immediately (up to 1 week) after the training or waiting period.
  Percentile ranks ranging from 0-100. Higher scores mean better outcome.
Behaviour Rating Inventory of Executive Function (BRIEF) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  T-scores ranging from 20 to 80 (M = 50, SD = 10). Higher scores mean better outcome.

OTHER OUTCOMES:
Physical Self-Description Questionnaire (PSDQ-S) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  Short version, Likert scale ranging from 1 to 6. Higher scores mean better outcome.
Conners-3 short form | At baseline
  T-scores ranging from 20 to 80 (M = 50, SD = 10). Higher scores mean better outcome.
Questionnaire for the Assessment of Resources and Competencies in Childhood and Adolescence (FRKJ) | At baseline; immediately (up to 1 week) after the training or waiting period; at 3-months follow-up.
  Stanine rank from 1-9. Higher score mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Regula Everts, Prof. Dr. phil., Principal Investigator — Division of Neuropaediatrics, Development and Rehabilitation, Department of Paediatrics, Inselspital, Bern University Hospital, University of Bern, Switzerland
Locations (1):
- Insespital, University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data can be shared upon reasonable request

REFERENCES:
- See also: Webpage MiA-study (german) — https://kinderklinik.insel.ch/de/lehre-und-forschung/forschung/forschung-nach-fachgebiet/neuropaediatrie/research-projects/mia-studie